CLINICAL TRIAL: NCT07120295
Title: Prospective Multicenter Clinical Performance Study of a Single-use Large Channel Digital Pancreaticobiliary Scope (DPS) With Compatible Accessories
Brief Title: Study of Large Channel Digital Pancreaticobiliary Scope (DPS) With Compatible Accessories
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Dragonfly Endoscopy Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-2548.cc; DGFLY-CLIN-2023-01 (Other: Dragonfly Endoscopy, Inc.)
Record Dates: First submitted 2025-04-30; First posted 2025-08-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Bile Duct Adenocarcinoma; Bile Duct Carcinoma
MeSH Terms: conditions — Bile Duct Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Interventional Group (Experimental)
  Interventions: Device: Dragonfly™ Digital Pancreaticobiliary System

INTERVENTIONS:
Device: Dragonfly™ Digital Pancreaticobiliary System — Dragonfly™ Digital Pancreaticobiliary System is indicated for use in the direct visualization of the biliary and pancreatic ducts for diagnostic and therapeutic interventions during endoscopic procedures. DPS is a single-use device that serves as an access and delivery catheter used with a proprietary DDC. The DDC is intended to control auto-illumination, and process images from the DPS for diagnostic and therapeutic applications during endoscopic procedures in the pancreaticobiliary system including the hepatic ducts.

SUMMARY:
This study plans to enroll up to 75 research subject who have a biliary disorder such as bile duct stones or intermediate biliary strictures. The purpose of this research is to assess whether the Dragonfly™ Pancreaticobiliary Scope functioned as intended in combination with the commercially available accessories during your scheduled endoscopy procedure. This includes achieving stone fragmentation of difficult biliary stone(s) while obtaining adequate tissue specimens for analysis. There will also be a Product performance evaluation as rated by the endoscopist operating the DPS System and evaluation of ergonomics and usability.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form;
2. Adult patients ≥ 21 years old;
3. Any patient who is required to undergo endoscopic retrograde cholangiopancreatography (ERCP) procedure with the clinical need to perform cholangioscopy for:

   1. Indeterminate biliary stricture, or
   2. Failed biliary stone extraction with conventional techniques.
4. Willing and able to follow study procedures and comply with study follow-up.

Exclusion Criteria:

1. Pregnancy or lactation;
2. Surgically or physiologically altered GI anatomy that precludes advancement of the duodenoscope for biliary cannulation;
3. Patients on anti-coagulants and anti-platelet medications that cannot be withheld pre-procedure, except for aspirin, 81mg;
4. Coagulopathy (INR > 1.8) or thrombocytopenia (Platelets < 50,000) that is not correctable and felt to be a contraindication to proceeding with biopsy or lithotripsy per the treating endoscopist;
5. Active suppurative cholangitis with evidence of purulent drainage at the time of papilla visualization;
6. Patients who are not candidates for anesthesia to permit ERCP.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Stone Fragmentation- Clearing of Biliary Stones | Up to 6 months
  Will evaluate the effectiveness of digital cholangioscopy (DC) in guiding fragmentation of difficult biliary stones. Will examine the efficacy of the intraductal lithotripsy procedure utilizing electrohydraulic lithotripsy in achieving biliary stone fragmentation and complete bile duct stone clearance among patients who have failed conventional stone extraction techniques. Stone fragmentation and complete ductal clearance will be assessed using descriptive statistics with interquartile range (IQR) for the number of procedures to achieve clearance at index or subsequent procedures. Ninety-five percent confidence intervals will be provided for descriptive statistics.
Tissue Acquisition during endoscopy procedure | Up to 6 months
  Will evaluate the ability of the DC to deliver tools to obtain adequate tissue samples (biopsies) to be analyzed for the presence or absence of disease, including cancer, infection, or other conditions in subjects with indeterminate strictures. Will use descriptive analysis with sensitivity, specificity, accuracy, median and IQR plus operating characteristics of visualization and sampling in those patients with indeterminate strictures. Will evaluate the diagnostic efficacy of the novel biopsy forceps in the context of indeterminate biliary strictures and provide robust evidence for clinical decision-making.

SECONDARY OUTCOMES:
Total procedure time | Up to 6 months
  Will evaluate the total procedure time for bile duct stones.
Product performance evaluation as rated by the endoscopist operating the DPS System | Up to 6 months
  Will evaluate the number of procedures required to achieve bile duct stone clearance after referral. Will summarize with descriptive statistics and report success rates. Ninety-five percent confidence intervals will be provided for descriptive statistics.
DPS Functionality during Endoscopy Procedures | Up to 6 months
  Will assess whether the DPS functioned as intended in combination with the commercially available accessories. Functioned as intended is defined as the ability to set up, provide visualization, deliver the accessory to the target location, use of the accessory according to the instructions for use. Will summarize with descriptive statistics and report success rates.
Ergonomics | Up to 6 months
  Will evaluate ergonomics by collecting anthropometric data from physician users. Will provide product performance evaluation data.
Lithotripsy fragmentation time | Up to 6 months
  Will evaluate lithotripsy fragmentation time for bile duct stones. Will summarize with descriptive statistics and report success rates.
Product Performance | Up to 6 months
  Will evaluate product performance for indeterminate biliary strictures as rated by the endoscopist operating the DPS system. Will summarize with descriptive statistics and report success rates.
Usability | At the completion of the study
  Will assess usability by the System Usability Scale. Will provide product performance evaluation data.
Visualization of biliary strictures | Up to 6 months
  Will evaluate the ability to adequately visualize biliary strictures, including the presence of both neoplastic (irregular nodular mucosa, irregular papillary projections, intraductal or villous mass, dilated and tortuous vessels with branching, infiltrative stricture, ulceration, and contact friability/ease of oozing) and benign (concentric, bandlike scar, uniform projections, thin vessels) characteristics. Will summarize with descriptive statistics and report success rates.
Visualization of stone or stricture characteristics | Up to 6 months
  Will evaluate usability by the ability to visualize stone or stricture characteristics as rated by the endoscopist operating the DPS system.
User satisfaction | At the completion of the study
  Will assess user satisfaction with the Net Promoter Score. Will provide product performance evaluation data.
Passing of device to target area | Up to 6 months
  Will evaluate usability by the ability to pass the lithotripsy device and/or stone removal device to the target area as rated by the endoscopist operating the DPS system.
Work | After each case
  Will assess the subjective assessment of work by the National Aeronautics and Space Administration-Task
Bile duct stone recurrence rate | At 6 months
  Will evaluate the bile duct stone recurrence rate. Will summarize with descriptive statistics and report success rates.

CONTACTS AND LOCATIONS:
Locations (1):
- Universtiy of Colorado Hospital, Aurora, Colorado, United States